CLINICAL TRIAL: NCT07088523
Title: Traditional Chinese Medicine Intervention for Ischemic Cardiovascular Disease Comorbid With Diabetes Mellitus: An Efficacy Comparative Study
Acronym: TICDEs
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0505604plus
Record Dates: First submitted 2025-07-06; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabete Mellitus; Ischemic Cardiovascular Disease
Keywords: Diabete Mellitus; Ischemic cardiovascular disease; real-world; Xintong Oral Liquid
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xintong TCM + Standard Treatment (Experimental): 1. Intensive phase: Xintong Oral Liquid 20 mL tid po, 4 weeks.
  2. Sequential phase: Xintong Oral Liquid 10 mL tid po, weeks 5-52.
  3. TCM decoction: Individualized herbal decoction based on TCM diagnosis (four diagnostic methods), administered for 14 days during intensive phase.
  Interventions: Drug: Xintong Oral Liquid (Sequential Phase); Drug: Xintong Oral Liquid (Intensive Phase); Drug: TCM Syndrome Differentiation Decoction
- Standard Treatment Only (Active Comparator): Guideline-based treatment for AMI with diabetes: aspirin (100 mg/day) + clopidogrel (75 mg/day) + atorvastatin (20 mg/day) + metformin (500 mg bid). Other antiplatelet/antidiabetic drugs may be added per clinician discretion.
  Interventions: Drug: Standard Treatment (Guideline-Based)

INTERVENTIONS:
Drug: Xintong Oral Liquid (Sequential Phase) — Xintong Oral Liquid (Lunan Pharmaceutical), 10 mL tid po from week 5 to 52.
  Arms: Xintong TCM + Standard Treatment
Drug: Xintong Oral Liquid (Intensive Phase) — Xintong Oral Liquid (Lunan Pharmaceutical), 20 mL tid po for 4 weeks.
  Arms: Xintong TCM + Standard Treatment
Drug: TCM Syndrome Differentiation Decoction — Individualized herbal decoction based on TCM diagnosis (four diagnostic methods), administered for 14 days during intensive phase.
  Arms: Xintong TCM + Standard Treatment
Drug: Standard Treatment (Guideline-Based) — Combination therapy including: 1. Antiplatelet: aspirin 100 mg/day + clopidogrel 75 mg/day. 2. Lipid-lowering: atorvastatin 20 mg/day. 3. Antidiabetic: metformin 500 mg bid (max 2000 mg/day). *Doses may be adjusted per local guidelines or patient tolerance.
  Arms: Standard Treatment Only

SUMMARY:
The population with comorbid ischemic cardiovascular disease (ICD) and diabetes mellitus (DM) has been growing rapidly, characterized by high mortality rates and frequent vascular event recurrence. DM exacerbates ischemic heart disease incidence and significantly elevates mortality in this comorbid population. Polypharmacy in these patients increases risks of adverse drug interactions and imposes substantial healthcare burdens. The pathological mechanisms of comorbidity demonstrate significant alignment with the TCM. Experimental studies indicate that Xintong Oral Liquid can ameliorate myocardial ischemia through multiple mechanisms to improve vascular endothelial function and microvascular dysfunction. This study aims to investigate the long-term effects of TCM intervention in patients with comorbid ICD and DM within 72 hours of symptom onset, and to evaluate whether the TCM treatment approach-centered on Xintong Oral Liquid within an integrated general treatment and syndrome differentiation framework-demonstrates superiority over control therapy in reducing 90-day major adverse cardiovascular and cerebrovascular events (MACCEs).

DETAILED DESCRIPTION:
This study is a large-scale, real-world, prospective, multi-center, non-randomized controlled clinical trail investigating the efficacy of a TCM therapeutic strategy with Xintong Oral Liquid as the core prescription in preventing major adverse cardiovascular and cerebrovascular events (MACCEs) in patients with Ischemic Cardiovascular Disease (ICD) complicated with Diabetes Mellitus (DM). This TCM therapeutic strategy is derived from the "toxins damaging collaterals" theory in TCM pathogenesis. All enrolled patients will receive standard treatment for ICD and DM based on the recommendations of guidelines. This study will employ natural selection grouping based on shared decision-making between physicians and patients, utilizing an open-label design with blinded endpoint assessment. An independent third-party endpoint adjudication committee will be established to conduct impartial evaluation and determination of all endpoint events. The study objective is to determine the following therapeutic effects of Xintong Oral Liquid as compared with standard treatment in the treatment of patients with ICD ccomplicated with DM: (1) 90-days incidence of the composite endpoints of major adverse cardiac and cerebrovascular events (MACCE), including cardiac death, myocardial re-infarction, emergent coronary revascularization and stroke; severe complications of STEMI (including cardiogenic shock, acute left heart failure, mechanical complications and malignant arrhythmias), in-stent thrombosis and major bleeding (Bleeding Academic Research Consortium [BARC] grade III and V); (2) Individual event of the 90-day primary endpoint; severe STEMI complications within 30-day treatment; target vessel failure (TVF) rate of PCI; MACCEs at 30, 180 and 365 days; follow-up assessments of SAQ-7 and EQ-5D-5L; the rate of readmission for heart failure; diabetic microangiopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years;
* Met the diagnostic criteria for myocardial infarction and type 2 diabetes mellitus;
* Within 72 hours of myocardial infarction onset;
* Met the diagnostic criteria of "toxins damaging collaterals"；
* Voluntary participation in the study with consent forms signed.

Exclusion Criteria:

* Long-term (>20 min) cardio-pulmonary resuscitation (CPR);
* Critical illness due to STEMI (such as serious cardiogenic shock, uncontrolled acute left heart failure or pulmonary edema, malignant arrhythmias, explicit mechanical complications, etc. );
* Suspected aortic dissection or acute pulmonary embolism;
* Bleeding history in any organ system within 1 month, or presence of active hemorrhage at any part of the body, or known hemorrhagic constitution, or severe coagulation disorder or current usage of anticoagulants;
* Uncontrolled severe diabetic ketoacidosis;
* Serious hepatic dysfunction or serious renal dysfunction ( ALT/AST≥3 ULN or eGFR<30mL/min/1.73 m2 or equiring dialysis );
* Serious COPD or respiratory failure;
* Severe infection (such as positive blood cultures, septic shock, and septic pneumonia, etc.);
* Neuropsychiatric system diseases or unconscious and unable to cooperate with examination and treatment;
* Malignancies or other conditions with expected survival time<1 year or unsuitability to participate in this study due to other diseases;
* Allergy to the ingredients of the research drugs;
* Women who are in pregnancy or nursery;
* Participation in clinical trial of other traditional Chinese medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4205 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
90-day Major Adverse Cardiovascular and Cerebrovascular Events (MACCEs) | 90 days
  Composite of: 1) Myocardial re-infarction (Third Universal Definition of MI); 2) Emergent coronary revascularization; 3) Stroke (NIHSS ≥1, imaging-confirmed); 4) Cardiovascular death (adjudicated by endpoint committee).

SECONDARY OUTCOMES:
30-day Severe STEMI Complications (Killip Class II-IV) | 30 days
  Composite of: 1) Cardiogenic shock (Killip IV); 2) Acute heart failure (Killip II-III); 3) Mechanical complications (e.g., ventricular septal rupture); 4) Malignant arrhythmia (sustained VT/VF). Assessed by adjudication committee.
30-day Severe Bleeding (BARC Type 3 or 5) | 30 days
  Bleeding Academic Research Consortium (BARC) criteria: Type 3 (overt bleeding with hemoglobin drop ≥3 g/dL or transfusion) or Type 5 (fatal bleeding).
365-day Target Vessel Failure (TVF) Rate | 365 days
  Composite of: 1) Cardiac death; 2) Target vessel myocardial infarction; 3) Target vessel revascularization (TVR). Angiographically confirmed by core lab.
Change in LVEF (%) from Baseline to 90 days | Baseline, 90 days
  Left ventricular ejection fraction measured by echocardiography (Simpson's biplane method).
Change in TyG Index from Baseline to 90 days | Baseline, 90 days
  Triglyceride-glucose index calculated as ln[fasting triglycerides (mg/dL) × fasting glucose (mg/dL)/2].
SAQ-7 Angina Frequency Score at baseline, 3, 6, 12 Months | Baseline, 3, 6, 12 Months
  Seattle Angina Questionnaire (SAQ-7) Domain 1 (Angina Frequency). Scale: 0-100 (higher=better).
EQ-5D-5L Utility Score at baseline, 3, 6, 12 Months | Baseline, 3, 6, 12 Months
  EuroQol 5-Dimension 5-Level (EQ-5D-5L) health-related quality of life. Scale: 0-1 (higher=better).
Heart Failure Readmission Rate at 180 Days and 365 Days | 180 days, 365 days
  Proportion of participants hospitalized for worsening heart failure (per modified Framingham criteria) within 180 days and 365 days post-treatment. Adjudicated by blinded Clinical Events Committee.

OTHER OUTCOMES:
Rate of Change in eGFR (mL/min/1.73 m²/year) | Baseline, 6 months, 12 months
  Estimated glomerular filtration rate (eGFR) calculated using CKD-EPI formula. Annualized rate of change derived from serial measurements at baseline, 6, and 12 months.
Rate of Change in UACR (mg/g/year) | Baseline, 6 months, 12 months
  Urine albumin-to-creatinine ratio (UACR) measured from first-morning void samples. Annualized rate of change calculated from baseline, 6, and 12-month data.
12-month Renal Composite Endpoint | 12 months
  Composite of: 1) Sustained ≥50% decline in eGFR from baseline; 2) Sustained eGFR <15 mL/min/1.73 m²; 3) Initiation of long-term dialysis or renal transplantation.
Change in Tubular Markers (α1-MG, β2-MG, NAG) at 12 Months | Baseline, 12 months
  Urinary biomarkers of tubular injury: α1-microglobulin (α1-MG), β2-microglobulin (β2-MG), and N-acetyl-β-D-glucosaminidase (NAG). Concentrations measured by immunoturbidimetry (α1-MG, β2-MG) and enzymatic assay (NAG).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Traditional Chinese Medicine Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) underlying the results of this study will not be shared publicly due to:
  1. Ethical and Legal Restrictions: The study involves sensitive health data of patients with acute myocardial infarction and diabetes, which are protected. Informed consent documents did not include provisions for public data sharing.
  2. Institutional Policies: Our institution's data governance framework requires that participant data be retained securely and used only for pre-specified research purposes.
  3. Practical Limitations: Anonymization of complex clinical datasets (e.g., including imaging, lab results, and follow-up records) cannot fully eliminate re-identification risks.
  Requests for de-identified data may be considered on a case-by-case basis for legitimate research purposes, subject to institutional review and data transfer agreements.